CLINICAL TRIAL: NCT04769921
Title: Full Arch Rehabilitations Through the Contemporary All-on-4 Concept
Acronym: AO4ContProt
Status: Active, not recruiting | Type: Observational
Sponsor: Malo Clinic (Other)
Collaborators: Nobel Biocare (Industry)
Responsible Party: Sponsor
Other Study IDs: AO4ContempProt
Record Dates: First submitted 2021-02-22; First posted 2021-02-25 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Edentulous Jaw
Keywords: All-on-4; All-on-four; dental implants; TiUltra; Xeal
MeSH Terms: conditions — Jaw, Edentulous | interventions — Dental Implants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- All-on-4 TiUltra and Xeal: Patients rehabilitated in the edentulous maxilla or mandible with an implant supported prosthesis through the All-on-4 Concept (2 anterior implants in the axial position and 2 posterior implants inserted with distal tilting). The implants used will be NobelParallel Conical Connection, with TiUltra surface. The abutments used will be Multi-unit abutments of internal connection with Xeal surface. The immediate prosthesis will be a high-density acrylic and 4 titanium cylinders. The definitive prosthesis will be a Titanium infrastructure with acrylic resin artificial gingiva and either acrylic or ceramic crowns.
  Interventions: Device: dental implants and abutments from Nobel Biocare

INTERVENTIONS:
Device: dental implants and abutments from Nobel Biocare — The implants will be inserted in an All-on-4 configuration; Abutments will be connected to the implants and serve as support for a full-arch implant-supported restoration.
  Other Names: NobelParallel Conical Connection; Multi-unit abutments with Xeal surface

SUMMARY:
It is necessary to generate more evidence on the outcome of contemporary protocols for full-arch rehabilitations supported by implants in immediate function in areas with limited quantity and density bone.

This research project aims to investigate the outcome of fixed prosthetic restorations supported by implants in immediate function for full-arch rehabilitation through the All-on-4 concept contemporary protocol, specifically: implant survival and success, prosthetic survival, marginal bone level and marginal bone level changes, soft tissue health parameters (Plaque index, Bleeding index, Pocket depth), incidence of biological and mechanical complications. A prospective cohort study design will be used in the investigation.

The sample of this study is estimated to consist in 43 patients rehabilitated with full-arch fixed prosthetic rehabilitations supported by implants in immediate function (All-on-4 concept) with 144 dental implants.

The cohort will be evaluated between baseline and 3 years of follow-up.

DETAILED DESCRIPTION:
Problem The fixed prosthetic rehabilitation through implants in immediate function is documented without prejudice of the outcome when compared to 2-stage surgery.1 One of the protocols for full-arch fixed prosthetic rehabilitation supported by implants in immediate function is the All-on-Four concept, which is documented with good long-term outcomes in both jaws.

Nevertheless, the protocols suffered a constant evolution throughout the 20 years of development of the All-on-4 concept. Evidence on the outcome full-arch rehabilitations supported by implants in immediate function through the All-n-4 concept contemporary protocol is needed. Therefore, the aim of this study was to document the rehabilitation of com¬pletely edentulous jaws through the contemporary All-on-4 concept rehabilitation protocol.

Objectives

* To evaluate the medium-term outcome (3 years) of full arch rehabilitations supported by implants in immediate function through the contemporary All-on-4 protocol
* To report the results

Study Endpoints Primary endpoint

* Prosthetic and implant survival over a 3-year follow-up period Secondary endpoint To evaluate Marginal Bone Level (MBL), Marginal Bone Level Changes 12, 24 and 36 months after procedure.
* To assess Soft tissue health parameters (Plaque index, Bleeding index, Pocket Depth)

Significance This investigation is important due to the need of studies reporting the outcome of full-arch rehabilitations supported by implants in immediate function through the All-on-4 concept contemporary protocol: Surgical Prosthetic and Maintenance.

Hypothesis The hypothesis to evaluate will be the distribution of survival, marginal bone resorption, incidence of biological and mechanical complications among the full-arch rehabilitations supported by implants in immediate function through the All-on-4 concept.

Materials and Methods Methodology This study will be performed at Maló Clinic in Lisbon. It is estimated to last for approximately 4 years.

The study design to be used will be a prospective single cohort study to evaluate the medium-term outcome of full-arch rehabilitations supported by implants in immediate function through the All-on-4 concept contemporary protocol (MALO CLINIC Protocol)2-4, composed of the Surgical, Prosthodontic and Maintenance protocols using dental implants and remaining prosthetic components from Nobel Biocare. A total of 36 subjects are planned to be included in the study over a recruitment period of 6 months.

The cohort will be evaluated between baseline and 3 years of function, regarding survival and clinical parameters established in this study.

There will be no risk for the participants, has the information will be collected using the standard of care during the implant maintenance appointment.

Population and Sample The population of this study consists in individuals eligible for full-arch rehabilitations with dental implants in immediate function through the All-on-4 concept, of both genders, without age restrictions, in any arch.

The sample of this study will consist in patients submitted to full-arch rehabilitations through the All-on-4 concept contemporary protocol.

Other inclusion criteria:

* Patients with enough bone quantity to be rehabilitated through the contemporary All-on-4 protocol using standard implants (7 to 25 mm of length);
* Patients that are interested in performing their follow-up and maintenance program at Maló Clinic);
* Patients that provide written informed consent to participate.

Exclusion criteria:

* Patients without enough bone quantity to be rehabilitated with the need of inserting zygomatic implants;
* Patients that exhibit bone graft reconstructions;

The selection of the participants to include the study group will be made after the evaluation of the inclusion and exclusion criteria.

Sample size The sample size is estimated to consist of 43 patients with a total of 172 dental implants inserted for full-arch rehabilitation through the All-on-4 concept contemporary protocol. The sample size calculation was based on a minimum number of 30 patients and considering a 30% dropout rate (n = 13 patients) during the study's three years of follow-up.

List and definition of variables:

Identification of the variable Definition of the variable (Dependent/Independent) Measured by:

Survival (implant and prosthetic) Dependent variable Nominal: 0: survival; 1: failure Marginal bone resorption Dependent variable Scale: measured through periapical radiographs, in millimeters between the implant shoulder and the most apical portion of implant-bone contact; difference between baseline, 1-year and 3-years measurements.

Biological complications Dependent variable Nominal: 0: absence; 1: presence Mechanical complications Dependent variable Nominal: 0: absence; 1: presence Patient age Independent variable Scale: number of years of life Patient gender Independent variable Nominal: 0:female; 1:male Smoking status Independent variable Nominal: 0:non-smoker; 1:smoker Systemic condition Independent variable Nominal: 0: absence; 1: presence Sub-classification according to the International Classification of Diseases, version 11.

Opposing dentition Independent variable Ordinal:

1. Fixed prosthesis over natural teeth
2. Implant supported prostheses
3. Miscellaneous
4. Natural teeth

External variables:

* Patients lost to follow-up;
* Patients withdrawing the study;
* The patient missing the control appointment;
* Interruption of the treatment by the patient;
* Patient deceased.

Clinical evaluation parameters:

The clinical parameters will be evaluated on the oral hygiene appointments at 10-days, 2 months, 4 months, 6 months, 1 year, 2 years and 3 years post-implant insertion.

* Success- determined according to the survival criteria developed by the authors;2
* Marginal bone resorption- Determined to the nearest 0.01 mm, by measuring the distance in mm from the implant shoulder to the first bone-implant interface. Digital periapical radiographs will be analyzed through software.

Sequence:

The sequence below represents the standard of care contemporary proceedings in a clinical maintenance appointment, listed with the exclusive objective of illustrating the clinical procedures regularly performed to collect clinical indexes (and not performed specifically for the execution of this study):

* Removal of fixed prosthetic rehabilitation;
* Evaluation of clinical parameters: Mobility, suppuration, plaque index, bleeding index, probing pocket depth;
* Evaluation of radiographic parameters: Marginal bone resorption;
* Implant maintenance and prophylaxis procedures;
* Reconnection of the fixed prosthetic rehabilitation.

Budget:

Item Amount (Eur) Description Dental implants, dental abutments, prosthetic cylinders, acrylic resin, acrylic resin teeth, titanium frameworks Waived by Nobel Biocare Necessary material to perform the implant-supported full-arch restorations.

Clinicians stipend Waived by Maló Clinic Full-time Clinicians stipend necessary to perform clinical evaluation of the implants during the follow-up of the study.

Study coordination Waived by Maló Clinic Study coordination during the follow-up of the study.

Statistical analysis Waived by Nobel Biocare Statistical analysis of the data collected during the study follow-up.

Radiographic analysis Waived by Nobel Biocare Radiographic evaluation at implant insertion, 1-year, 2-year and 3-year follow-up.

Production, publication and reporting the study outcomes Waived by Maló Clinic Production of report; submission to publication in peer-reviewed journal; Report study results.

Total 0 €

Statistical analysis:

In this study, the data will be treated by means of descriptive and inferential statistics.

The data will be treated using the SPSS software version 25.0 (SPSS Inc., Chicago, IL, USA).

Implant and prosthetic survival will be computed through life tables. Marginal bone loss will be evaluated using descriptive statistics: average values with 95% confidence intervals and standard deviations will be reported.

The incidence of biological, mechanical and prosthetic complications will be evaluated using descriptive statistics (frequencies).

Adverse events:

An adverse event is defined as any undesirable clinical occurrence in a subject whether it is considered to be device related or not. If the adverse event is regarded as device related it is stated as an adverse device effect.

An adverse event or adverse device effect may be serious\severe or non-serious\non-severe. If, as result of an adverse event during a clinical investigation, a subject has to be hospitalized, or their hospitalization is unduly prolonged due to potential disability or danger to life due to an intervention has been required or the event is terminal, the adverse event or adverse effect is regarded as serious.

All serious adverse events must be reported to the Ethic Committee without any delay.

Ethical aspects:

This investigation will be carried out in accordance to the ethical principles and guidelines stated in the Declaration of Helsinki.

The Investigation should be evaluated and approved by a Local Ethical Committee prior to including the first subject in the investigation. The application to the Ethic Committee is to be made by the responsible investigators.

The patients' data will be registered in a computer database, using a code system. This means that the identity of each subject will be unknown to the investigators. The patients' medical records and radiographs will be used exclusively for data collection. No extra interventions for study purposes will be performed to any patient. No recalls will be performed at any time with the intention of specifically collecting information from the patients.

It is also of great importance that each subject receives oral and written information about the investigation, and that she/he must only participate if they truly want to do so. Also, the subjects must be aware of the fact that they can withdraw from the investigation at any time and for any reason without jeopardizing their future treatment.

Furthermore, the subjects should be made aware of the fact that the data from his/her treatment will be registered in a computer database, but that she/he will only be registered through a code system. This means that the identity of each subject will be unknown to all others than the doctor performing the treatment. Each subject is entitled to take part of the information stored about her/his treatment. This information is to be handed out by the treating doctor.

For more information on subject information, consent and data, please see Appendix 2.

Database management:

The data collected from the forms will be introduced in a digital database (Microsoft Office Excel 2003®). The database management will be the responsibility of the Malo Clinic.

Monitoring Monitoring will be carried out by the Ethical Committee. The investigator will issue a final report that will be distributed.

Archiving the documents The data will be archived by the Malo Clinic and will be kept for 8 years after the completion of the study. After this time, the digital database will be erased.

ELIGIBILITY:
Inclusion Criteria:

* Patients with enough bone quantity to be rehabilitated through the contemporary All-on-4 protocol using standard implants (7 to 25 mm of length);
* Patients that are interested in performing their follow-up and maintenance program at Maló Clinic);
* Patients that provide written informed consent to participate.

Exclusion Criteria:

* Patients without enough bone quantity to be rehabilitated with the need of inserting zygomatic implants;
* Patients that exhibit bone graft reconstructions;
* Hindrance to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population of this study consists in individuals eligible for full-arch rehabilitations with dental implants in immediate function through the All-on-4 concept, of both genders, without age restrictions, in any arch.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2019-02-19 (Actual); Primary Completion 2022-07-08 (Actual); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Prosthetic survival | annually up to 3 years of follow-up
  Survival of the implant-supported prosthesis at the end of the follow-up period
Dental implants survival | annually up to 3 years of follow-up
  Survival of the dental implants at the end of the follow-up period

SECONDARY OUTCOMES:
Marginal bone loss | 1-, 2- and 3-years
  Evaluation of marginal bone loss by comparing bone levels at evaluation points with baseline (day of surgery)
Plaque index | 1-, 2- and 3-years
  Evaluation of the modified Plaque Index at designated time points
Bleeding index | 1-, 2- and 3-years
  Evaluation of the modified Bleeding Index at designated time points
Probing pocket depts | 1-, 2- and 3-years
  Evaluation of the probing pocket depths in millimeters in 4 points on each implant and recoded in "</ 4 mm" and "> 4 mm"

OTHER OUTCOMES:
Biological complications | During the 3 years of follow-up
  Evaluation of the incidence of biological complications (abcess, fistula, infection, peri-implant pathology) during the follow-up of the study.
Mechanical complications | During the 3 years of follow-up
  Evaluation of the incidence of mechanical complications (loosening or fracture of any prosthetic component) during the follow-up of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Miguel A de Araújo Nobre, PhD, Study Chair — Malo Clinic
Locations (1):
- Malo Clinic, Lisbon, Lisbon District, Portugal

IPD SHARING:
Plan to Share IPD: No